CLINICAL TRIAL: NCT02979249
Title: Effect of Oral Iron Therapy on Erythrocyte Protoporphyrin Levels in the Erythropoietic Protoporphyrias
Brief Title: Oral Iron for Erythropoietic Protoporphyrias
Acronym: EPP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Manisha C Balwani, Associate Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 08-0959-1001; U54DK083909 (NIH)
Record Dates: First submitted 2016-11-29; First posted 2016-12-01 (Estimated); Results first posted 2020-09-11 (Actual); Last update posted 2020-09-11 (Actual); Status verified 2020-08

CONDITIONS: Erythropoietic Protoporphyria; EPP; X-linked Protoporphyria; XLP
Keywords: Interventional; open-label; EPP; XLP; porphyria
MeSH Terms: conditions — Protoporphyria, Erythropoietic; Protoporphyria, Erythropoietic, X-Linked Dominant; Porphyrias | interventions — Iron

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oral Iron (Experimental): standard dose of iron pills
  Interventions: Drug: Oral Iron

INTERVENTIONS:
Drug: Oral Iron — for one year
  Other Names: Ferrous sulfate USP

SUMMARY:
In the medical literature there are conflicting reports on whether iron improves symptoms in patients with EPP and XLP. Giving iron to people who are iron deficient is thought to improve EPP symptoms. However, this has never been systematically tested. Therefore, the purpose of this study is to determine the effect of oral iron for EPP and XLP patients.

DETAILED DESCRIPTION:
This is a clinical trial, which means its purpose is to study an intervention or treatment. In this study all patients with EPP or XLP will be given a standard dose of iron pills and monitored for one year. There is currently no effective Food and Drug Administration (FDA) approved treatment for EPP or XLP in the US. Giving iron to patients with low ferritin (a measure of body iron stores) levels may help improve their EPP symptoms by decreasing erythrocyte protoporphyrin levels.

Patients will be asked come to the study site once every three months over the course of a year for a total of five visits. At these visits the study doctors will check in with participants and some blood and urine samples will be taken. Participants will not be charged for any of the lab tests that are being done for part of this study alone. In between these study visits there will be phone call to check in and see how participants are doing. All patients in this study will receive iron pills at no cost to them.

ELIGIBILITY:
Inclusion Criteria:

* Enrollment in the Longitudinal Study of the Porphyrias
* Male or female age ≥18 years
* History of nonblistering cutaneous photosensitivity
* Biochemical findings - A marked increase in erythrocyte protoporphyrin (total erythrocyte protoporphyrin >400 ug/dL) with a predominance of metal-free protoporphyrin
* Serum ferritin ≤30 ng/mL at baseline
* Able to tolerate oral iron

Exclusion Criteria:

* History of liver or bone marrow transplant or clinically significant liver dysfunction as determined by the investigator
* Known or suspected allergy to oral iron based on patient report
* Clinical evidence of active and ongoing GI bleeding
* Use of any other clinical or experimental therapy in the past 3 months
* Individuals with elevations of porphyrins in plasma or erythrocytes due to other diseases (i.e. secondary porphyrinemia) such as liver and bone marrow diseases
* Patients with any clinically significant comorbid conditions, which in the opinion of the investigator, precludes participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-12; Primary Completion 2019-07-19 (Actual); Study Completion 2019-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Manisha Balwani, MD, MS, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (6):
- United States (6):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - University of California, San Francisco, California
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Texas Medical Branch, Galveston, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Derived] Balwani M, Naik H, Overbey JR, Bonkovsky HL, Bissell DM, Wang B, Phillips JD, Desnick RJ, Anderson KE. A pilot study of oral iron therapy in erythropoietic protoporphyria and X-linked protoporphyria. Mol Genet Metab Rep. 2022 Nov 14;33:100939. doi: 10.1016/j.ymgmr.2022.100939. eCollection 2022 Dec. PMID 36406817
- See also: Porphyrias Consortium website — https://www.rarediseasesnetwork.org/cms/porphyrias/Studies

RESULTS

PARTICIPANT FLOW:
Groups:
- Oral Iron: standard dose of oral iron pills for one year
Period: Overall Study
Arm/Group | Oral Iron
Started | 16
Completed | 10
Not Completed | 6
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 4

BASELINE CHARACTERISTICS:
Arm/Group | Oral Iron
Number analyzed (Participants) | 16
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.8 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Erythrocyte Protoporphyrin Levels
Description: Relative difference in erythrocyte protoporphyrin levels between baseline and 12 months after treatment
Time Frame: Baseline and at 12 months
Measure: Mean (Standard Deviation); unit: µg/dL
Arm/Group | Oral Iron
Number analyzed (Participants) | 10
µg/dL
  Baseline | 2314.6 (1820.3)
  12 months | 2240.4 (2312.6)

2. Secondary Outcome: Mean Change in EPP-specific Quality of Life Questionnaire
Description: Quality of life tool designed to capture the specific issues that patients with EPP experience. Score range is 0-100, higher scores represent higher levels or satisfaction, lower scores represent more impacted quality of life. Mean change at 12 months as compared to baseline.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: mean change in score on a scale
Arm/Group | Oral Iron
Number analyzed (Participants) | 10
mean change in score on a scale | 3.3 (18.3)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Oral Iron
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Iron (N=10)
Diarrhea (Gastrointestinal disorders) | 1
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 1
Conjunctivitis (Eye disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Oral Iron (N=10)
Abdominal Pain (Gastrointestinal disorders) | 2
Photosensitivity (Skin and subcutaneous tissue disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Sinusitis (Infections and infestations) | 1
Dyspepsia (Gastrointestinal disorders) | 1
Elevated Protoporphyrin (Metabolism and nutrition disorders) | 1 — greater than 35% of baseline
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Urinary Tract Pain (Renal and urinary disorders) | 1
Elevated Protoporphyrin (Blood and lymphatic system disorders) | 1 — greater than 35% of baseline
Mucosal Infection (Infections and infestations) | 1
Constipation (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-14): https://cdn.clinicaltrials.gov/large-docs/49/NCT02979249/Prot_SAP_000.pdf